## Official Title of the Study:

Twelve-Month Short-Term Marginal Bone Remodeling at Monolithic Zirconia Full-Arch Prostheses in the Maxilla and Mandible: A Clinical Study

#### **NCT Number:**

NCT: Not yet assigned

# **Document Type:**

Study Protocol

**Document Date:** July 9, 2020

#### **Version:**

1.0

## **Sponsor:**

Universitat Internacional de Catalunya (UIC)

Principal Investigator: Luis Carlos Garza Garza

## **Study Sites:**

Universitat Internacional de Catalunya

#### **Study Information**

Study Number: REST-ECL-2020-02

Principal Investigator: Luis Carlos Garza Garza

Co-Investigators: Ricardo David Palacios, Eduardo Crooke De Aguilar

Supervisor: Miguel Roig

**Department:** Restorative and Esthetic Dentistry

Research Line: Basic and applied research in dentistry

### **Participant Consent Statement**

| I, Mr./Ms.: |
|-------------|

- I have received verbal information about the study and I have read the written information attached, of which I have been given a copy.
- I understand what has been explained to me.
- I have been able to discuss the study and ask questions to the responsible professional.
- I give my consent to participate in the study and I understand that my participation is entirely voluntary.
- I understand that I may withdraw from the study at any time without this affecting my future medical care.

By signing this informed consent form, I authorize my personal data to be used as described in this document and in compliance with the applicable data protection regulations.

I understand that I will receive a copy of this informed consent form.

| Signatures |
|------------------------------------------------|
| Signature of the patient ID / Passport Number: |
| Date of signature |